CLINICAL TRIAL: NCT01223716
Title: Does Video Game Play Induce Plasticity in the Visual System of Adults With Amblyopia?
Brief Title: An Active Approach to Treat Amblyopia: Video Game Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Roger Winghong Li, Research Specialist, University of California, Berkeley
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CPHS#2003-11-83; R01EY001728 (NIH)
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Amblyopia
Keywords: amblyopia treatment; neural plasticity; perceptual learning; vision therapy; spatial vision; video games; occlusion therapy
MeSH Terms: conditions — Amblyopia | interventions — Crossing Over, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perceptual learning (Experimental)
  Interventions: Behavioral: Perceptual learning
- Video Game (Experimental)
  Interventions: Behavioral: Video Game
- Occlusion Therapy (Experimental)
  Interventions: Behavioral: Crossover (Occlusion therapy + Video Game)

INTERVENTIONS:
Behavioral: Perceptual learning — Research participants will be asked to practice a visual discrimination task (e.g. position acuity, contrast sensitivity, stereoacuity etc) in our laboratory for a period of time (2 hrs/day, 5 days/week).
  Other Names: vision therapy; vision training
  Arms: Perceptual learning
Behavioral: Video Game — Research participants will be asked to play "off-the-shelf" video games in our laboratory for a period of time (2 hrs/day, 5 days/week).
  Other Names: vision therapy; vision training
  Arms: Video Game
Behavioral: Crossover (Occlusion therapy + Video Game) — Phase 1. Research participants will be required to cover the good eye during the day in order to push the brain to use the amblyopic eye (2 hrs/day, 5 days/week for 2-4 weeks).
  Phase 2. Research participants will be required to cover the good eye during the day in order to push the brain to use the amblyopic eye (2 hrs/day, 5 days/week for 2-4 weeks).
  Other Names: vision therapy; vision training
  Arms: Occlusion Therapy

SUMMARY:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. This study uses psychophysical measures to study neural plasticity in adults with amblyopia.

DETAILED DESCRIPTION:
Amblyopia, a developmental abnormality that impairs spatial vision, is a major cause of vision loss, resulting in reduced visual acuity and reduced sensitivity to contrast. Our previous findings (see CITATIONS) show that the adult amblyopic brain is still plastic and malleable, suggesting that active approach is potential useful in treating amblyopia. The goal of this project is to assess the limits and mechanisms of neural plasticity in amblyopic spatial vision. This study uses psychophysical measures to study neural plasticity in adults with amblyopia. Research participants will be asked to play video games with the amblyopic eye for a period of time. A range of visual functions will be monitored during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults with amblyopia (Age >15 years)
* Amblyopia: interocular visual acuity difference of at least 0.1 logMAR
* All forms of amblyopia: Strabismic, anisometropic, refractive, deprivative, meridional amblyopia

Exclusion Criteria:

* Any ocular pathological conditions (eg macula abnormalities, glaucoma), nystagmus

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Amblyopic vision | 9 months
  Improvement in amblyopic vision : visual acuity and stereoacuity

SECONDARY OUTCOMES:
Spatial vision | 9 months
  Improvement in spatial vision (positional acuity and spatial attention)
Temporal vision | 9 months
  Improvement in temporal processing and temporal vision (attentional blink)

CONTACTS AND LOCATIONS:
Overall Officials: Roger W Li, OD, PhD, Principal Investigator — School of Optometry, Univeristy of california-Berkeley; Dennis M Levi, OD, PhD, Principal Investigator — School of Optometry, Univerisity of California-Berkeley
Locations (1):
- Minor Hall 486, School of Optometry, University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li RW, Provost A, Levi DM. Extended perceptual learning results in substantial recovery of positional acuity and visual acuity in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2007 Nov;48(11):5046-51. doi: 10.1167/iovs.07-0324. PMID 17962456
- [Background] Li RW, Young KG, Hoenig P, Levi DM. Perceptual learning improves visual performance in juvenile amblyopia. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3161-8. doi: 10.1167/iovs.05-0286. PMID 16123415
- [Background] Li RW, Levi DM. Characterizing the mechanisms of improvement for position discrimination in adult amblyopia. J Vis. 2004 Jun 1;4(6):476-87. doi: 10.1167/4.6.7. PMID 15330715
- [Background] Chung ST, Li RW, Levi DM. Identification of contrast-defined letters benefits from perceptual learning in adults with amblyopia. Vision Res. 2006 Oct;46(22):3853-61. doi: 10.1016/j.visres.2006.06.014. Epub 2006 Aug 22. PMID 16930666
- [Background] Chung ST, Kumar G, Li RW, Levi DM. Characteristics of fixational eye movements in amblyopia: Limitations on fixation stability and acuity? Vision Res. 2015 Sep;114:87-99. doi: 10.1016/j.visres.2015.01.016. Epub 2015 Feb 7. PMID 25668775
- [Result] Li RW, Klein SA, Levi DM. Prolonged perceptual learning of positional acuity in adult amblyopia: perceptual template retuning dynamics. J Neurosci. 2008 Dec 24;28(52):14223-9. doi: 10.1523/JNEUROSCI.4271-08.2008. PMID 19109504
- [Result] Chung ST, Li RW, Levi DM. Learning to identify near-threshold luminance-defined and contrast-defined letters in observers with amblyopia. Vision Res. 2008 Dec;48(27):2739-50. doi: 10.1016/j.visres.2008.09.009. Epub 2008 Oct 18. PMID 18824189
- [Result] Levi DM, Li RW. Improving the performance of the amblyopic visual system. Philos Trans R Soc Lond B Biol Sci. 2009 Feb 12;364(1515):399-407. doi: 10.1098/rstb.2008.0203. PMID 19008199
- [Result] Levi DM, Li RW. Perceptual learning as a potential treatment for amblyopia: a mini-review. Vision Res. 2009 Oct;49(21):2535-49. doi: 10.1016/j.visres.2009.02.010. Epub 2009 Feb 27. PMID 19250947
- [Result] Li RW, Tran TT, Craven AP, Leung TW, Chat SW, Levi DM. Sharpening coarse-to-fine stereo vision by perceptual learning: asymmetric transfer across the spatial frequency spectrum. R Soc Open Sci. 2016 Jan 20;3(1):150523. doi: 10.1098/rsos.150523. eCollection 2016 Jan. PMID 26909178
- [Result] Li RW, Ngo CV, Levi DM. Relieving the attentional blink in the amblyopic brain with video games. Sci Rep. 2015 Feb 26;5:8483. doi: 10.1038/srep08483. PMID 25715870
- [Result] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514
- [Result] Chung ST, Li RW, Levi DM. Learning to identify near-acuity letters, either with or without flankers, results in improved letter size and spacing limits in adults with amblyopia. PLoS One. 2012;7(4):e35829. doi: 10.1371/journal.pone.0035829. Epub 2012 Apr 30. PMID 22558234